CLINICAL TRIAL: NCT03596268
Title: Functional Imaging Reserve in NeuroHIV
Acronym: FIRN
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Missouri, St. Louis (Other); Temple University (Other); University of California, San Diego (Other)
Responsible Party: Sponsor
Other Study IDs: 201805047
Record Dates: First submitted 2018-07-09; First posted 2018-07-23 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: HIV
MeSH Terms: interventions — Diagnostic Imaging; Spinal Puncture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Biospecimen Retention: Samples With DNA — Blood (plasma and cellular) and CSF will be obtained for assessment of immune dysfunction (immune activation and exhaustion). Blood and CSF will be stored on ice until centrifuged (within 30 minutes of collection). EDTA-coagulated blood will be used to isolate PBMCs using the standard Ficoll separation method. PBMCs will be frozen at -80C in 90% FBS 10% RPMI for flow cytometry phenotypic analyses. Plasma, CSF and PBMCs will be aliquoted into vials and frozen (-80C) until at least 60 participants have completed their visit, at which time samples will be sent and batch-analyzed by Dr. Burdo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Persons Living with HIV (PLWH): Persons 20-80 years old with a documented HIV infection for at least 1 year, who are on a stable cART medication regimen for at least 1 year, and have an undetectable plasma HIV RNA (<50 copies/ml).
  Interventions: Diagnostic Test: Imaging; Diagnostic Test: Serum Laboratory Tests; Diagnostic Test: Lumbar Puncture
- HIV- Controls: Persons 20-80 years old with confirmed HIV- status matched to PLWH cohort with similar age, sex, education, and race.
  Interventions: Diagnostic Test: Imaging; Diagnostic Test: Serum Laboratory Tests; Diagnostic Test: Lumbar Puncture

INTERVENTIONS:
Diagnostic Test: Imaging — 3T Prisma MRI
Diagnostic Test: Serum Laboratory Tests — Blood (plasma and cellular) will be collected.
Diagnostic Test: Lumbar Puncture — CSF will be collected

SUMMARY:
The purpose of this research study is to look at the brain's efficiency and ability to make up for deficits in the front of the brain to see if people living with HIV (PLWH) are still able to perform well on various cognitive tasks even though there are other underlying processes at work, like inflammation, that affect the brain in a negative way. Results of this study may provide insight into the pathophysiology of disease and may reveal arenas for future possible interventions in PLWH who have impaired neuropsychological performance.

DETAILED DESCRIPTION:
This proposal systematically characterizes brain efficiency and recruitment in virologically suppressed persons living with HIV (PLWH) and demographically similar HIV uninfected (HIV-) controls. This proposal collects advanced functional neuroimaging that provide critical information about cerebral blood flow (CBF) and brain connectivity (functional connectivity strength; FCS); quantitative measures of immune dysfunction in the blood and cerebrospinal fluid (CSF) (immune activation and immune exhaustion); and neuropsychological performance testing. This overall goal of this proposal is to delineate the interplay between dysfunction in frontal networks and recruitment of compensatory networks that underlie the neuropsychiatric symptoms seen in PLWH.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 80 years old
* documented HIV infection for at least 1 year or confirmed HIV - status
* PLWH must be on stable cART regimen for at least 12 months with undetectable plasma HIV RNA (less than 50 copies per mL)
* at least 9 years of education
* able to provide informed consent
* if female, a negative pregnancy test and not breast feeding
* able to undergo an MRI scan

Exclusion Criteria:

* significant neurological disorders (e.g. stroke, head injury with loss of consciousness for more than 5 minutes, developmental learning disability)
* active uncontrolled Axis I psychiatric disorder according to the DSM 5
* current or history of substance use disorder (including, but not limited to amphetamines, cocaine, alcohol, opiates, and barbiturates)
* prescribed blood thinners
* allergic to lidocaine or similar anesthetic
* history of any bleeding disorder
* contraindication to MRI scanning (e.g. claustrophobia, pacemaker, etc.)
* pregnant or breastfeeding

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult persons living with HIV (PLWH) and demographically similar healthy HIV- controls
Sampling Method: Non-Probability Sample
Enrollment: 284 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Brain Efficiency and Recruitment - Determine the neuroimaging signatures of brain efficiency and recruitment in virologically suppressed PLWH. | 5 years
  The investigators will compare the recruitment of compensatory networks between the PLWH and HIV- controls using multiple linear regression. In exploratory analyses the investigators will compare the brain efficiency between PLWH and HIV-, using similar multiple regression models, controlling for confounders. Among PLWH, the investigators will study the association of brain efficiency with neuropsychological performance testing using multiple regression models.

SECONDARY OUTCOMES:
Effects of Aging - Determine the effects of aging on brain efficiency and recruitment in virologically suppressed PLWH. | 5 years
  The investigators will compare the recruitment (response) between the four HIV age groups (HIV- <50 year old, HIV- ≥50 years old, HIV+ <50 years old, and HIV+ ≥50 years old) using a multiple regression (ANCOVA) model, adjusting for potential confounders (age, sex, education, past substance use, and CVD). The pairwise comparisons of primary interest is between the HIV- <50 years old and the HIV- ≥50 years old groups. Among the PLWH only, the investigators will compare the brain efficiency r (response) between the younger and older group using multiple regression, adjusting for potential confounders. Secondly, a mediation analysis will examine the role of immune dysfunction (activation and exhaustion) markers as mediators of this relationship.

CONTACTS AND LOCATIONS:
Overall Officials: Beau M Ances, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data might be shared when the study has closed.

DOCUMENTS (1):
  • Informed Consent Form (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT03596268/ICF_001.pdf